CLINICAL TRIAL: NCT03511950
Title: The Relationship Between the Change of Resting Energy Expenditure(REE) and Nutritional Status in Peritoneal Dialysis(PD) Patients With Peritonitis.
Brief Title: The Relationship Between the Change of Resting Energy Expenditure and Nutritional Status .
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor in Renal Division, Department of Medicine, Peking University First Hospital
Other Study IDs: REE and peritonitis
Record Dates: First submitted 2018-04-01; First posted 2018-04-30 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Peritonitis; Resting Energy Expenditure; Nutrition
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peritonitis is a common and devastating complication in patients on peritoneal dialysis (PD). It is a known fact that persistent inflammatory state and nutritional deterioration are closely associated with increased mortality in PD patients.And resting energy expenditure(REE) is significantly increased in acute and chronic inflammation in patients with chronic kidney disease (including dialysis patients).However,it is limited to the changing trend and duration of REE in peritonitis.Investigators hypothesize that the increase in total energy consumption resulting from the increase of REE which may accompany with decreased energy intake will lead to negative energy balance and nutritional deterioration, which may affect the prognosis of patients.Therefore,a prospective cohort study will be designed to dynamically research the change of REE accompanied with the nutrition status in peritonitis and provide the basis for peritonitis management in the future.

ELIGIBILITY:
Inclusion Criteria:

* Receiving PD for>3 months
* Age between 18 and 80 years
* Confirm diagnosis of peritonitis

Exclusion Criteria:

* Disability
* Other acute complications: including systemic infections except for peritonitis, acute cardia-cerebrovascular disease in one month
* Active hepatitis and musculoskeletal diseases in the past
* Cancer and is treated with chemoradiotherapy within 1 year
* Severe edema of the whole body or a large amount of body cavity effusion
* Thyroid dysfunction
* History of hormonal drugs use
* During pregnancy or lactation
* Mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients with confirm diagnosis of peritonitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The relationship between the change of REE and the change of albumin | 90 days
  Method: REE, indirect calorimetry

SECONDARY OUTCOMES:
The relationship between the change of REE and the change of BMI | 90 days
  The relationship between the change of REE and the change of BMI during 90 days after peritonitis
The relationship between the change of REE and the change of handgrip strength | 90 days
  The relationship between the change of REE and the change of handgrip strength during 90 days after peritonitis
The relationship between the change of REE and the change of Fat mass | 90 days
  Method: REE, indirect calorimetry; Fat mass, Bioelectrical impedance
The relationship between the change of REE and the change of lean body mass | 90 days
  Method: REE, indirect calorimetry; lean body mass, Bioelectrical impedance

OTHER OUTCOMES:
The relationship between the change of REE and the outcome of patients | 90 days or 180days
  outcome including death and transfer to hemodialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China